CLINICAL TRIAL: NCT05362604
Title: Top Benefits of the Prenatal Diagnosis of the Fetal Esophageal or Intestinal Atresia
Brief Title: Prenatal Diagnosis of the Fetal Esophageal or Intestinal Atresia
Acronym: DANATRESIA
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DANATRESIA
Record Dates: First submitted 2022-02-08; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-02

CONDITIONS: Antenatal Management of the Fetal Gastrointestinal Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prenatal: patients affected by confirmed fetal esophageal, duodenal or intestinal atresia and followed in our high-risk pregnancy unit, and scheduled for delivery between 38 and 39 weeks in our tertiary center, regardless of the patient's place of residence
  Interventions: Procedure: scheduled delivery at a tertiary center
- postnatal: patients with unsuspected fetal atresia who delivered in their local hospitals: their newborns were transferred to our tertiary hospital within 24 hours and the mother had the option to be also transferred in order to follow her baby.

INTERVENTIONS:
Procedure: scheduled delivery at a tertiary center — Neonatal units in French hospitals are classified in three levels. The intention is for infants requiring high level care to receive it in a tertiary neonatal unit within the same network when appropriate. In case of known fetal gastro-intestinal artesia, the prenatal care includes obstetric consultation and level 3 ultrasound scheduled every four weeks at our unit until the end of the pregnancy, antenatal consultations with a specialized multidisciplinary team, and an antenatal visit of the birth center to reduce the parental anxiety.
  Groups: prenatal

SUMMARY:
Aim- to investigate how prenatal diagnosis of fetal esophageal or intestinal atresia impacts obstetric and neonatal outcomes.

Methods- This was a retrospective cohort study at a single center. The study population comprised 51 consecutive pregnancies, including 29 mothers (57%) and their fetuses affected by prenatally diagnosed fetal esophageal or intestinal atresia, and 22 mothers (43%) and their babies with postnatally diagnosed fetal esophageal or intestinal atresia.

DETAILED DESCRIPTION:
Aim- to investigate how prenatal diagnosis of fetal esophageal or intestinal atresia impacts obstetric and neonatal outcomes.

Methods- This was a retrospective cohort study at a single center. The study population comprised 51 consecutive participants, including 29 mothers (57%) and their fetuses affected by prenatally diagnosed fetal esophageal or intestinal atresia, and 22 mothers (43%) and their babies with postnatally diagnosed fetal esophageal or intestinal atresia.

ELIGIBILITY:
Inclusion Criteria:

* all pregnancies affected by fetal esophageal, duodenal or intestinal atresia referred to our prenatal diagnosis unit
* all newborns managed for such atresia in our unit of pediatric surgery

Exclusion Criteria:

* termination of pregnancy,
* stillbirth,
* the false positive cases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 51 mother-baby pairs
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
gestational age of delivery | 1 year
  weeks
mode of delivery | 1 year
  Vaginal, Operative vaginal, Elective cesarean section, Cesarean section for fetal indication

SECONDARY OUTCOMES:
neonatal morbidity | 1 year
  Age at surgery, Cutaneous stoma, Anastomotic leakage, Mechanical ventilation, Phototherapy, Infection
length of hospital stay | 1 year
  Length of neonatal intensive care unit stay, Length of neonatal reanimation stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No